CLINICAL TRIAL: NCT03058783
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Study to Evaluate the Efficacy and Safety of IDP-124 Lotion for the Treatment of Moderate to Severe Atopic Dermatitis in Pediatric and Adult Subjects
Brief Title: Efficacy and Safety of IDP-124 Lotion for the Treatment of Moderate to Severe Atopic Dermatitis in Pediatric and Adult Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-124A-302
Record Dates: First submitted 2016-12-21; First posted 2017-02-23 (Actual); Results first posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDP-124 Lotion (Experimental): IDP-124 Lotion, twice-daily application
  Interventions: Drug: IDP-124 Lotion
- IDP-124 Vehicle Lotion (Active Comparator): IDP-124 Vehicle Lotion, twice-daily application
  Interventions: Drug: IDP-124 Vehicle Lotion

INTERVENTIONS:
Drug: IDP-124 Lotion — IDP-124 Lotion, twice-daily application
  Arms: IDP-124 Lotion
Drug: IDP-124 Vehicle Lotion — IDP-124 Vehicle Lotion, twice-daily application
  Arms: IDP-124 Vehicle Lotion

SUMMARY:
Efficacy and Safety of IDP-124 Lotion for the Treatment of Moderate to Severe Atopic Dermatitis in Pediatric and Adult Subjects

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Study to Evaluate the Efficacy and Safety of IDP-124 Lotion for the Treatment of Moderate to Severe Atopic Dermatitis in Pediatric and Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 2 years of age and older
* Written and verbal informed consent must be obtained; subjects less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if subject reaches age of consent during the study they should be re-consented at the next study visit)
* Nonimmunocompromized male or female who failed to respond adequately to other topical prescription treatment for AD or for whom those treatments are not advisable
* Subjects must be willing to comply with study instructions and return to the clinic for required visits; subjects under the age of consent must be accompanied by the parent or legal guardian at the time of assent/consent signing

Exclusion Criteria:

* Females who are pregnant, breast feeding, or who wish to become pregnant during the study period
* Active cutaneous bacterial or viral infection in any treatment area at Baseline (eg, clinically infected AD)
* Sunburn, extensive scarring, or pigmented lesion(s) in any treatment area at Baseline, which would interfere with evaluations
* History of confounding skin conditions, eg, psoriasis, rosacea, erythroderma, or ichthyosis (other than ichthyosis vulgaris)
* History or presence of:
* basal cell carcinoma of skin effectively treated more than 2 years ago
* carcinoma of cervix effectively treated more than 5 years ago
* immunological deficiencies or diseases, HIV, or serious recurrent infection
* clinically significant severe renal insufficiency or severe hepatic disorders
* Current or recent serious infection

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Valeant Pharmaceitucals
Locations (1):
- Valeant Site 05, Fremont, California, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDP-124 Lotion | IDP-124 Vehicle Lotion
Started | 216 | 110
Completed | 180 | 80
Not Completed | 36 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-124 Lotion | IDP-124 Vehicle Lotion | Total
Number analyzed (Participants) | 216 | 110 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (20.21) | 33.1 (20.46) | 31.8 (20.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 54 | 176
  Male | 94 | 56 | 150
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 23 | 13 | 36
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 69 | 34 | 103
  White | 110 | 59 | 169
  More than one race | 9 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had at Least a 2-grade Reduction From Baseline at Week 6 in the Investigator Global Assessment (IGA) Scale and Had an IGA at Week 6 That Equated to "Clear" or "Almost Clear"
Description: Investigator Global Assessment (IGA) was determined based on evaluator-blinded evaluations of the inflammatory signs of atopic dermatitis. Evaluations were scored using a 5-point scale from clear (0) to severe (4), with higher numbers indicating worse scores.
Time Frame: Baseline to Week 6
Measure: Number; unit: percentage of participants
Arm/Group | IDP-124 Lotion | IDP-124 Vehicle Lotion
Number analyzed (Participants) | 216 | 110
percentage of participants | 42.04 | 32.73

2. Secondary Outcome: Percentage of Participants Who Had at Least a 2-grade Reduction From Baseline in the Investigator Global Assessment (IGA) Scale and Had an IGA That Equated to "Clear" or "Almost Clear"
Description: as for outcome 1
Time Frame: Baseline to Week 10
Measure: Number; unit: percentage of participants
Arm/Group | IDP-124 Lotion | IDP-124 Vehicle Lotion
Number analyzed (Participants) | 216 | 110
percentage of participants
  Week 2 | 18.89 | 8.73
  Week 4 | 28.70 | 24.91
  Week 10 | 31.67 | 29.64

3. Secondary Outcome: Percentage of Participants Who Had Eczema Area Severity Index (EASI) 75
Description: EASI 75 is defined as at least a 75% reduction in the Eczema Area Severity Index (EASI) score from Baseline. EASI is composite score based on the evaluated severity of 4 key signs of AD (i.e., erythema, infiltration/papulation, excoriation and lichenification), and the extent of disease in each of the 4 body regions (i.e., head/neck, trunk, upper limbs, and lower limbs). The area of involvement (affected by inflammation, not including dry skin) of each of the 4 body regions is determined and represented by a numeric coded value based on a scale from 0 to 6. The 4 body regions are assessed separately for each sign/symptom, and the average degree of severity of each sign in each of the 4 body parts is assigned a score of 0 (none) to 3 (severe) on a scale that allows half-unit increments. The EASI score ranges from 0 to 72, with higher scores being worse.
Time Frame: Baseline to Week 10
Measure: Number; unit: percentage of participants
Arm/Group | IDP-124 Lotion | IDP-124 Vehicle Lotion
Number analyzed (Participants) | 216 | 110
percentage of participants
  Week 4 | 33.61 | 26.18
  Week 6 | 46.11 | 37.45
  Week 10 | 43.24 | 34.00

4. Secondary Outcome: Percentage of Participants Who Had at Least a 1 Grade Improvement From Baseline in the Severity of Pruritus Score and a Pruritus Score Equating to "None" or "Mild"
Description: Pruritis was assessed on a 4-point scale with 0 (none) to 3 (severe) and higher scores being worse.
Time Frame: Baseline to Week 2
Measure: Number; unit: percentage of participants
Arm/Group | IDP-124 Lotion | IDP-124 Vehicle Lotion
Number analyzed (Participants) | 216 | 110
percentage of participants
  Week 1 | 46.19 | 37.41
  Week 2 | 52.76 | 39.81

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | IDP-124 Lotion | IDP-124 Vehicle Lotion
All-Cause Mortality (participants affected / at risk) | 0/216 | 0/110
Serious Adverse Events (participants affected / at risk) | 2/216 | 0/110
Other Adverse Events (participants affected / at risk) | 0/216 | 0/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-124 Lotion (N=216) | IDP-124 Vehicle Lotion (N=110)
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT03058783/Prot_SAP_000.pdf